CLINICAL TRIAL: NCT06812195
Title: Plate Over Humeral Nail in Deformity Correction of Femur in Adult Osteoporotic Bone
Brief Title: Periprosthetic Plate Over Humeral Nail
Acronym: osteoporosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, Lecturer of orthopedics, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPON; PPOND (Other: Faculty of Medicine for Girls Al-Azhar University)
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Osteopenia, Osteoporosis
Keywords: deformity; osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Congenital Abnormalities; Osteoporosis | interventions — Bone Plates

STUDY DESIGN:
Intervention Model Description: Under spinal anesthesia in supine position, lateral approach to the femur is used to do corrective osteotomies and introduction of humeral nail according to preoperative plan. After that, plate is applied to lateral border to the feoral shaft. Weight bearing is allowed after confirmation of union after 6 weeks. Regular visits every 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- plate over humeral nail (Experimental): spinal anesthesia in supine position, lateral approach to the femur is used to do corrective osteotomies and introduction of nail according to preoperative plan. After that, plate is applied to lateral border to the feoral shaft
  Interventions: Device: Plate and nail

INTERVENTIONS:
Device: Plate and nail — spinal anesthesia in supine position, lateral approach to the femur is used to do corrective osteotomies and introduction of nail according to preoperative plan. After that, plate is applied to lateral border to the femoral shaft

SUMMARY:
use of plate over humeral nail in deformity correction of femur in adult osteoporotic bone

DETAILED DESCRIPTION:
small IM interlocking nail, such as humeral nail, could be used in femoral fixation in normal adolescent patients due to the advantages of the entry point lateral to tip of greater trochanter resulting in avoiding iatrogenic vascular injury and being the IM locking device with smaller diameter and shorter length than conventional femoral nail which was appropriate for small-sized adolescent femoral anatom

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic bone with femoral deformity.
* Osteogenesis imperfecta. --Vitamin D deficiency ricket

Exclusion Criteria:

* Uncooperative patient.

  -- Skeletally immature
* Not receiving medical treatment.
* Patient with history of allergy to drugs used in the study.
* Neuromuscular pathology, previous trauma, or surgery to the leg

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Metal failure | 2 years
  Number of cases with bending or protrusion

CONTACTS AND LOCATIONS:
Overall Officials: Hesham M Elbaseet, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon JE, Khanna N, Luhmann SJ, Dobbs MB, Ortman MR, Schoenecker PL. Intramedullary nailing of femoral fractures in children through the lateral aspect of the greater trochanter using a modified rigid humeral intramedullary nail: preliminary results of a new technique in 15 children. J Orthop Trauma. 2004 Aug;18(7):416-22; discussion 423-4. doi: 10.1097/00005131-200408000-00004. PMID 15289686